CLINICAL TRIAL: NCT02857374
Title: Intravital Microscopy (IVM) During Sentinel Lymph Node (SLN) Biopsy for Melanoma
Brief Title: Intravital Microscopy in Identifying Tumor Vessels in Patients With Stage IB-IIIC Melanoma Undergoing Sentinel Lymph Node Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I 284116; NCI-2016-01076 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 284116 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2016-07-29; First posted 2016-08-05 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Stage IB Skin Melanoma; Stage IIA Skin Melanoma; Stage IIB Skin Melanoma; Stage IIC Skin Melanoma; Stage IIIA Skin Melanoma; Stage IIIB Skin Melanoma; Stage IIIC Skin Melanoma
MeSH Terms: conditions — Melanoma | interventions — Fluorescein; Fluoresceins; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (intravital microscopy) (Experimental): Patients receive indocyanine green and fluorescein sodium injection IV and then undergo intravital microscopic observation over 15-20 minutes during standard of care sentinel node biopsy.
  Interventions: Procedure: Diagnostic Microscopy; Drug: Fluorescein Sodium Injection; Other: Laboratory Biomarker Analysis; Procedure: Sentinel Lymph Node Biopsy

INTERVENTIONS:
Procedure: Diagnostic Microscopy — Undergo intravital microscopy
Drug: Fluorescein Sodium Injection — Given IV
  Other Names: AK-Fluor; Fluorescite
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Sentinel Lymph Node Biopsy — Undergo standard of care sentinel node biopsy
  Other Names: Sentinel Node Biopsy; Sentinel node biopsy alone; SLNB; SNB

SUMMARY:
This pilot clinical trial studies intravital microscopy in identifying tumor vessels in patients with stage IB-IIIC melanoma undergoing sentinel lymph node biopsy. By examining sentinel lymph nodes through intravital microscopy before they are removed, doctors may learn specific information regarding how melanoma may spread to lymph nodes and other sites of the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of intravital microscopy in characterizing the microvasculature of the sentinel lymph node (SLN) in melanoma patients requiring SLN biopsy.

SECONDARY OBJECTIVES:

I. To identify vascular blood flow parameters and flow kinetics associated with the sentinel lymph node vasculature and define the utility of using commonly used fluorescent agents during human intravital microscopy and correlate with clinical outcomes (time to recurrence, survival), as a potential basis for a novel prognostic tool and/or microstaging technique.

TERTIARY OBJECTIVES:

I. To determine the relationship between live microscopically-recorded images and pathology slides in terms of vessel density and vessel diameter.

OUTLINE:

Patients receive indocyanine green and fluorescein sodium injection intravenously (IV) and then undergo intravital microscopic observation over 15-20 minutes during standard of care sentinel node biopsy.

After completion of study treatment, patients are followed up at 3 weeks and then every 6 months for 5 years or every 3 months for 2 years and every 6 months for another 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Melanoma tumor that meets indications for a groin SLN biopsy with a >= 10% risk of having metastasis to the draining lymph node (i.e. stage IB to stage IIIC melanoma of the lower body below the umbilicus)
* Participant must be eligible for a groin sentinel lymph node (SLN) biopsy
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Sentinel lymph node is deemed inaccessible to microscopic observation during the operative procedure (i.e. sentinel node maps to a deep location or area outside of the groin)
* Renal dysfunction as defined as creatinine clearance < 70 mL/min by Cockroft-Gault equation
* Any known allergy or prior reaction to fluorescein, indocyanine green, iodine, or shellfish
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to undergo observational study (may also include preoperative testing results including electrocardiogram [EKG], chest x-ray, or pulmonary function tests)
* Any condition that excludes SLN biopsy as the standard of care (e.g. lymphadenectomy indicated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Feasibility of intravital microscopy in characterizing the microvasculature of the SLN in melanoma determined by successful visualization of at least 6 of 10 patients during Part I | Up to 3 weeks
  The visualization method will be deemed successful in patients with tumor vessel identification, measurement of tumor vessel diameters, determining vessel density, and visualizing fluorescein/indocyanine green within the tumor vessels.

SECONDARY OUTCOMES:
Flow kinetics associated with the sentinel lymph node vasculature | Up to 5 years
  Sample sentinel lymph node characteristics obtained from the intervention will be characterized using descriptive statistics (means, medians) and 95% confidence intervals.
Survival | Up to 5 years
  Assessed using Kaplan Meier and Proportional Hazards methods. Collected through routine follow-up processes.
Time to progression | Up to 5 years
  Assessed using Kaplan Meier and Proportional Hazards methods. Collected through routine follow-up processes.
Treatment response | Up to 5 years
  Assessed using Logistic Regression. Collected through routine follow-up processes.
Utility of using commonly used fluorescent agents during human intravital microscopy | Up to 3 weeks
Vascular blood flow parameters associated with the sentinel lymph node vasculature | Up to 5 years
  Sample sentinel lymph node characteristics obtained from the intervention will be characterized using descriptive statistics (means, medians) and 95% confidence intervals.

OTHER OUTCOMES:
Blood vessel density and diameter assessed from live microscopically-recorded images and from pathology slides | Up to 5 years
  The relationship between the live microscopically-recorded images and the pathology slides in terms of vessel density and vessel diameter will be determined. Correlations between microscopic observations (vessel diameter, density, blood flow velocity, vessel hierarchy tissue penetration of fluorescein/indocyanine green) with pathologic node positivity and clinical outcomes (time to recurrence, survival) will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Skitzki, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States